

Study Number & Rev.: IRB Protocol CL-006

**Identifiers:** NCT03469128

Study Title: Cognitive Processing Therapy Versus Sertraline for the Treatment of Comorbid

Substance Use Disorder and Post-Traumatic Stress Disorder in Egyptian patients

**Study Design:** Randomized clinical trial

**Sponsor Name:** The British University in Egypt

Sponsor Address: El-Sherouk City, Cairo, Egypt

**Data Analysis:** 01-01-2016

**Expected Completion Date:** December 2019

Principal Investigator: Dr. Amani Elbarazi, Clinical Practice Department, Faculty of

Pharmacy, The British University in Egypt, P.O. Box 43, El-Sherouk

City, Cairo 11837, Egypt

## STATEMENT OF CONFIDENTIALITY

The information contained herein is confidential information that is the sole and exclusive property of The British University in Egypt and may not be divulged to any person (except as required by law) without the prior written consent of The British University in Egypt.

## Protocol signature page

The undersigned has read and understood the trial protocol detailed above and agrees to conduct the trial in compliance with the protocol.

| Dr. Amani Elbarazi | Amani | BUE3570 | 01-01-2016 |
|------------------------|-----------|-----------------|------------|
| Principal Investigator | Signature | Site name or ID | Date |
| (Please print name) | | number | |



| Fac | culty | of F | haı | rmacy |
|------|---------|------|-----|----------|
| _ــة | بدلــــ | الص | ـبة | <u> </u> |

## **Consent Form**

Project: Cognitive Processing Therapy Versus Sertraline for the Treatment of Comorbid Substance Use Disorder and Post-Traumatic Stress Disorder in Egyptian patients

| Principal investigator: Amani | Elbarazi | | |
|---|---|---|---|
| 1- I confirm that I have read and the above study and had the to ask questions. | | | |
| 2- I understand that my participation is voluntary and that I am free to withdraw at any time, without giving any reason and without my treatment being affected. | | | |
| 3- In the case of withdrawal I understand that any information collected up to that point can still be used by the researchers | | | |
| 4- I agree to take part in study p of assessments and filling of | | re that this involves answeringssessments on paper copies. | ng a set |
| 5- I agree to supply the research GP/ Consultant. These details | | ils and those of my | |
| Name of Participant | Date | Signature | |
| Researcher<br>Dr. Amani Elbarazi | Date<br> | Signature | |
| Please supply your GP/Consulta | | | |
| Address: | | | |
| | ••••• | | |

MANY THANKS FOR AGREEING TO TAKE PART IN THIS STUDY.